CLINICAL TRIAL: NCT06526637
Title: User Testing of the Palliate Intervention, Supporting Lay Carers to Prepare and Administer Anticipatory Medications to Loved Ones at Home at the End of Life.
Brief Title: User Testing of an End of Life Medication Support Intervention for Lay Carers (Palliate).
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Oak Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OFIL-20-279
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: End of Life; Support, Family
Keywords: Palliative Care
MeSH Terms: conditions — Death | interventions — myotrophin

STUDY DESIGN:
Intervention Model Description: The study will use direct observational methods in a workshop setting. Participants will be randomised to receive one of three Palliate training and material versions. Randomisation will be completed ahead of study commencement using a random number generator to allow the researcher time to prepare and set up the selected training information and materials. Randomisation will be conducted in blocks of three to ensure an even number randomised to each of the study arms (intervention version 1,2 and 3).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Version 1 of Palliate (Active Comparator): Participants will be randomised to receive this version of Palliate training and materials.
  Interventions: Other: Paper Package
- Version 2 of Palliate (Experimental): Participants will be randomised to receive this version of Palliate training and materials.
  Interventions: Other: V1 + Preparation Sheet
- Version 3 of Palliate (Experimental): Participants will be randomised to receive this version of Palliate training and materials.
  Interventions: Other: V2 + Video Training

INTERVENTIONS:
Other: Paper Package — Paper based (as per current practice at Central and North West London (CNWL) NHS Foundation Trust) version of Palliate.
  Arms: Version 1 of Palliate
Other: V1 + Preparation Sheet — Paper based version of Palliate plus a preparation sheet, that provides visual cues as to what equipment is required for the preparation and administration of the medications.
  Arms: Version 2 of Palliate
Other: V2 + Video Training — Hybrid - paper based materials, preparation sheet, and video instructions available via an interactive portable document format (PDF) version of the training materials.
  Arms: Version 3 of Palliate

SUMMARY:
The aim of this study is to evaluate the acceptability, safety and efficiency of the Palliate intervention.

The Palliate intervention is a nurse-led process that includes training and documentation materials to support lay carers in administering top up medications to loved ones at the end of life at home. The Palliate intervention was designed based on the CARiAD* intervention using user testing and has been successfully piloted and rolled out in Central and North West London National Health Service (NHS) Foundation Trust.

*CARer-ADministration of as-needed sub-cutaneous medication for breakthrough symptoms in homebased dying patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older and able to communicate in English.

Exclusion Criteria:

* Individuals aged less than 18 years old and/or unable to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Acceptability | Through study completion per participant (≤ 5 weeks)
  Participant scores of acceptability of the intervention as per the responses on the Theoretical Framework of Acceptability (TFA) questionnaire. Free text or verbal responses noted when completing the questionnaire will be thematically analysed as informed by the TFA.
  The TFA questionnaire is an eight-item questionnaire. Raw total scores range from 8 (the worst possible score) to 40 (the best possible score).

SECONDARY OUTCOMES:
Usability | Through study completion per participant (≤ 5 weeks)
  Participant scores of usability as per the System Usability Scale (SUS) questionnaire.
  The SUS is a ten-item attitude Likert scale giving a global view of subjective assessments of usability. Scores range from 0 (the worst possible score) to 100 (the best possible score).
Incidence of error | Through study completion per participant (≤ 5 weeks)
  Medication Error will be defined as any of the following - Wrong medication
  Wrong dose - if >10% deviation from the prescribed dose.
  Wrong indication - was the selected medication and dose correct for the symptoms presented.
  Administration error - incorrect process of administration
  Documentation error - failure to document or incorrect documentation.
  (Wrong patient- n/a, Wrong route- n/a, Wrong concentration- n/a, Wrong diluent- n/a)
Efficiency | Through study completion per participant (≤ 5 weeks)
  Time taken to prepare and administer each medication. This will be defined as - Start = the moment the participant begins reading the scenario Finish = the moment the medication has been administered Time for documentation will also be recorded.
Factors contributing to error, potential errors and acceptability of the intervention | Through study completion per participant (≤ 5 weeks)
  Hierarchical Task Analysis - The workflow of reading the scenario, through to preparation, administration and documentation of the medications will be micro-analysed and mapped. Medication events that are found to be erroneous, take longer than anticipated or deem to be problematic by the participant or researcher/s will be analysed against the workflow map to identify which step in the process was the likely cause of the issue.
Learnability/ Retained learning | Through study completion per participant (≤ 5 weeks)
  Differences in the incidence of error and time to complete task between a, each medication preparation and administration and b, between the first and second visit.
Actual and perceived barriers and opportunities from the participants regarding the use of the Palliate intervention | Through study completion per participant (≤ 5 weeks)
  Guided by the theoretical framework of acceptability- Short semi-structure interviewers following participation in the user testing. And/or completion of a questionnaire with a combination of open and closed questions.

CONTACTS AND LOCATIONS:
Overall Officials: Leila Shepherd, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No